CLINICAL TRIAL: NCT05409417
Title: Exploratory Study on Combined Conversion Immunotherapy for Liver Metastasis of MSS Type Initial Unresectable Colorectal Cancer Based on Gene Status
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2022058
Record Dates: First submitted 2022-01-03; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drugs, Investigational; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab Combined With chemotherapy (Experimental): Tislelizumab Combined With XELOX and Bevacizumab or Tislelizumab Combined With FOLFOX and Cetuximab
  Interventions: Drug: Experimental drug

INTERVENTIONS:
Drug: Experimental drug — Tilelizumab combined with XELOX and bevacizumab or tislelizumab combined with FOLFOX and cetuximab
  Other Names: Tilelizumab combined with chemotherapy

SUMMARY:
Evaluation of tislellimab combined with XELOX and bevacizumab or tislelizumab combined with FOLFOX and cetuximab regimen in patients with liver metastases from colorectal cancer Rate and R0 resection rate and safety.

ELIGIBILITY:
Inclusion Criteria:

3.1 Entry criteria:

1. Male or female, age ≥18 years old, ≤75 years old
2. Liver metastases of colorectal adenocarcinoma confirmed by histology, liver metastases are initially unresectable
3. RAS gene mutation or wild type, BRAF wild type, MSS type
4. ECOG physical status is 0 to 1 points
5. Life expectancy is at least 12 weeks
6. Absolute neutrophil count (ANC)>1.5×109/L, hemoglobin>8g/dL and platelets>100×109/L (based on the normal value of the clinical trial center)
7. Prothrombin time (PT) <1.5 times the upper limit of normal and normal thromboplastin time (APTT) <1.5 times the upper limit of normal
8. Laboratory examination, serum creatinine is less than or equal to 1.5 times the upper limit of the reference range of normal value (if serum creatinine rises, 24-hour urine must be collected, except for those with 24-hour creatinine clearance> 50ml/min)
9. When there is no liver metastasis, ALT or AST is less than or equal to 2.5 times the upper limit of the normal value reference range, and serum total bilirubin is less than or equal to 1.5 times the upper limit of the normal value reference range; for patients with liver metastases, ALT or AST is less than Or equal to 5 times the upper limit of the reference range of normal values, and serum total bilirubin is less than or equal to 3 times the upper limit of the reference range of normal values
10. Women of childbearing age must be willing to adopt adequate contraceptive measures during study drug treatment
11. Signed informed consent
12. According to the definition of RECIST 1.1, the investigator determines that the patient has a measurable disease. Tumor lesions located in the area of previous radiotherapy are considered measurable if they are confirmed to have progressed.

Exclusion Criteria:

3.2 Exclusion criteria:

1. An active autoimmune disease that requires systemic treatment (i.e., use of disease-relieving drugs, corticosteroids, or immunosuppressive agents) occurred in the previous 2 years. Replacement therapies (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments.
2. Diagnosed with immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first administration of the experimental treatment. After consultation with the sponsor, the use of physiological doses of corticosteroids may be approved.
3. Anti-tumor monoclonal antibody (mAb) received within 4 weeks before the first day of the study, or adverse events caused by the drug received 4 weeks before have not yet recovered (ie ≤ grade 1 or reach baseline level).
4. Have received chemotherapy, targeted small molecule therapy or radiotherapy within 2 weeks before the first day of the study, or the adverse events caused by the previously received drugs have not yet recovered (ie ≤ grade 1 or reach the baseline level). Note: Subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 hair loss are exceptions to this standard and may be eligible to participate in the study. a. If subjects have undergone major surgery, they must fully recover from the toxicity and/or complications caused by the intervention before starting treatment.
5. Other malignant tumors are known to be progressing or requiring active treatment. Exclude skin basal cell carcinoma, skin squamous cell carcinoma or cervical carcinoma in situ that have received radical treatment.
6. Active central nervous system (CNS) metastasis and/or cancerous meningitis are known to exist. Subjects who have received brain metastasis therapy can also participate in this study, provided that their condition is stable (no disease progression confirmed by imaging examination at least 4 weeks before the first administration of the trial treatment, and all neurological symptoms have returned to Baseline level), there is no evidence that new or enlarged brain metastases have occurred, and steroid therapy should be discontinued at least 7 days before the first dose of the trial treatment. This exception does not include cancerous meningitis, which should be excluded regardless of whether the clinical condition is stable. Have a history of pneumonia (non-infectious) requiring steroid treatment or are currently suffering from pneumonia (non-infectious).
7. Active infections requiring systemic treatment.
8. It is possible to confuse the test results, prevent the subjects from participating in the research in the whole process of medical history or disease evidence, abnormal treatment or laboratory values, or the researcher believes that participating in the research is not in the subjects' best interests.
9. It is known that there are mental or drug abuse diseases that may affect compliance with the test requirements.
10. During pregnancy or lactation, or expected to be during the planned trial period (from the beginning of the screening visit to 120 days after the last dose of the study treatment (applicable to the Pembrolizumab group), or until 180 days after the last dose of the study treatment ( Applicable to paclitaxel group)) conceived female subjects, or male subjects whose spouse becomes pregnant.
11. Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibody) infection.
12. Known to have active hepatitis B or C. Active hepatitis B is defined as a known positive result of HBsAg and an HBV viral load exceeding 2000 IU/ml (104 copies/ml). Active hepatitis C is defined as a known hepatitis C antibody positive, and the quantitative result of known hepatitis C RNA is higher than the detection limit of the analytical method. Note: HCV RNA (quantitative) and HBsAg testing will be performed during the screening period; if there are results obtained within 3 months before the screening period, it can also be used.
13. Live vaccines have been vaccinated within 30 days before the planned start date of the study treatment. a. Note: Seasonal influenza vaccines for injection are generally inactivated influenza vaccines and are allowed to be used; but intranasal influenza vaccines (such as FluMist®) are live attenuated vaccines and are not allowed.
14. BRAF gene mutation type, MSI-H

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Conversion rates | 3 months
  Conversion rates based on RECIST1.1
R0 resection rate | 3 months
  R0 resection rate based on RECIST1.1
Drug Safety | 12 months
  Drug safety assessed by CTCAE v4.0; Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

SECONDARY OUTCOMES:
ORR | 3 months
  objective response rate based on RECIST1.1
PFS | through study completion，an average of 2 years
  Progression-Free Survival %
OS | through study completion，an average of 3 years
  Overall survival %
DCR | through study completion，an average of 2 years
  Disease control rate % based on RECIST1.1

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes